CLINICAL TRIAL: NCT02592330
Title: Safety and Feasibility of Cultivated Autologous Limbal Epithelial Cell Transplantation in the Treatment of Limbal Stem Cell Deficiency (LSCD)
Brief Title: Limbal Stem Cell Deficiency (LSCD) Treatment With Cultivated Stem Cell (CALEC) Graft
Acronym: CALEC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ula Jurkunas, Associate Professor, Harvard Medical School, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-124H
Record Dates: First submitted 2015-02-09; First posted 2015-10-30 (Estimated); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: LSCD treatment; Limbal Stem Cell Deficiency; CALEC; Cultivated Autologous Limbal Epithelial Cell Transplantation; Corneal epithelial stem cells; Corneal scarring; Corneal opacity; Chemical injury eye; Thermal injury eye; Autologous stem cell; Epithelial defect; Corneal cloudiness; Ocular burn; Ocular injury; Autograft; Conjunctival Limbal Autograft; LSCD research; Chronic contact lens wear; Chronic keratoconjunctivitis; Corneal conjunctivalization; Corneal fibrovascular pannus; Corneal neovascularization; Corneal regeneration; Infectious keratitis; Limbal epithelial stem cell deficiency; Ocular injury drug toxicity; Ocular surface disorder; Neovascularization pannus; Neurotrophic keratitis; Ocular surface Inflammation; Eye injury ionizing radiation; Eye injury ultraviolet radiation; Corneal pannus; Corneal wound healing; Neurotrophic keratopathy; LSCD trial; Stem cell therapy; Epithelial surface integrity; Regrowing corneas
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Corneal Injuries; Corneal Opacity; Eye Injuries; Corneal Neovascularization

STUDY DESIGN:
Intervention Model Description: All subjects will receive the study intervention, a stem cell graft cultivated from their own cells.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cultivated Autologous Limbal Epithelial Cell (CALEC) graft (Experimental): Participants will have a corneal biopsy in their non-diseased eye, which will provide cells for the creation of the CALEC graft. The CALEC will be made at the Good Manufacturing Practice (GMP) Laboratory, Dana Farber Cancer Institute and transported to Mass. Eye and Ear Infirmary for application to the participant's diseased eye during their standard corneal reconstruction procedure.
  Interventions: Procedure: Biopsy to collect limbal epithelial stem cells that will be cultivated into a graft; Biological: Cultivation of Limbal epithelial cells into a graft; Procedure: CALEC Transplant

INTERVENTIONS:
Procedure: Biopsy to collect limbal epithelial stem cells that will be cultivated into a graft — Cultivated autologous limbal epithelial cell (CALEC) therapy utilizes a bio-engineered composite of ex vivo expanded autologous corneal epithelial cells and an FDA-approved amniotic membrane (AmnioGraft®, Bio-Tissue, Inc.) to reconstruct the ocular surface. A small biopsy (2-3 mm2) from the patient's contralateral eye serves as a source epithelial (stem) cells that are expanded on the amniotic membrane in culture and the resulting product is surgically transplanted onto the cornea after excision of the fibrovascular pannus.
  Other Names: Cultivated Autologous Limbal Epithelial Cell (CALEC)
Biological: Cultivation of Limbal epithelial cells into a graft — A graft is manufactured for transplant
Procedure: CALEC Transplant — Limbal epithelial cells are obtained from the healthy fellow eye and cultivated in a lab for later transplantation into the diseased eye.
  Other Names: Conjunctival Limbal Autograft

SUMMARY:
The main aim of the study is to determine the safety and feasibility of a cultivated autologous limbal epithelial cell (CALEC) transplantation in the treatment of limbal stem cell deficiency.

DETAILED DESCRIPTION:
This is an open label, single center study to assess safety, feasibility, and efficacy of Cultivated Autologous Limbal Epithelial Cell (CALEC) grafts in 17 patients with unilateral limbal stem cell deficiency (LSCD).

Participants will have a corneal biopsy in their non-diseased eye, which will provide cells for the creation of the CALEC graft. The CALEC will be made at the Good Manufacturing Practice (GMP) Laboratory, Dana Farber Cancer Institute and transported to Mass. Eye and Ear Infirmary for application to the participant's diseased eye during their standard corneal reconstruction procedure. Subjects will be monitored up to month 18 post-transplant to assess for any delayed adverse events of the product (CALEC) or procedure as well as assessment of the durability of the transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants age 18 to <90 years old at time of enrollment
* Ability of a subject or guardian/legal representative to provide written informed consent and to comply with study assessments for the full duration of the study.
* Patients with unilateral limbal stem cell deficiency (LSCD) as determined by conjunctivalization of the cornea defined by fibrovascular pannus more than 2 mm from the limbus for greater than or equal to 6 clock hours.
* Additional optional criteria:

  * Lack of limbal palisades of Vogt for greater than or equal to 9 clock hours
  * Goblet cell presence as defined by impression cytologic criteria

Exclusion Criteria:

* Corneal or ocular surface infection within 30 days prior to study entry or CALEC transplantation
* Ocular surface malignancy
* Uncontrolled diabetes with most recent HgA1c greater than 8.5%
* Renal Failure with eGFR below 60 mL/min per 1.73 m2
* Aspartate aminotransferase and alanine aminotransferase levels greater than 3 times institutional upper limit of normal
* Total bilirubin greater than 2 times institutional upper limit of normal (except patients with known Gilbert's syndrome)
* Platelet levels less than 100,000 or greater than 450,000 per microliter
* Hemoglobin levels of less than 11.0 g/dL in men or less than 10.0 g/dL in women
* Prothrombin time greater than 16 seconds and activated partial thromboplastin time greater than 35 seconds in patients not taking warfarin and an international normalized ratio greater than 3 in patients taking warfarin
* Inability to tolerate monitored anesthesia
* HIV infection or AIDS
* Active Hepatitis B or C
* Pregnancy (positive test) or lactation
* Participation in another simultaneous medical investigation or trial
* Severe cicatricial eye disease
* Severe dry eye disease as determined by Schirmer's test less than 1mm in at least one eye.
* Any medical, psychiatric, debilitating disease/disorder or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.
* Signs of current infection, including fever and current treatment with antibiotics.
* History of allo-limbal transplantation
* Presence of allergy to the CALEC graft or any of the chemical components within its formulation.

Exclusion Based on Donor Eye:

* Conjunctivalization of the cornea defined by fibrovascular pannus more than 2 mm from the limbus for greater than or equal to 3 clock hours
* Lack of limbal palisades of Vogt for greater than or equal to 3 clock hours
* History of allo-limbal transplantation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ula Jurkunas, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yavuz Saricay L, Kaufman AR, Johns LK, Yin J, Samarakoon L, Ayala AR, Maguire M, Parekh M, Hernandez Rodriguez DE, Daley H, Dana R, Armant M, Ritz J, Jurkunas UV. Central Cornea Changes on Anterior Segment OCT and In Vivo Confocal Microscopy After Autologous Limbal Epithelial Cell Transplantation. Cornea. 2025 Mar 28. doi: 10.1097/ICO.0000000000003865. Online ahead of print. PMID 40152603
- [Derived] Jurkunas UV, Kaufman AR, Yin J, Ayala A, Maguire M, Samarakoon L, Johns LK, Parekh M, Li S, Gauthier A, Negre H, Shaw KL, Hernandez Rodriguez DE, Daley H, Dana R, Armant M, Ritz J. Cultivated autologous limbal epithelial cell (CALEC) transplantation for limbal tem cell deficiency: a phase I/II clinical trial of the first xenobiotic-free, serum-free, antibiotic-free manufacturing protocol developed in the US. Nat Commun. 2025 Mar 4;16(1):1607. doi: 10.1038/s41467-025-56461-1. PMID 40038272

RESULTS

PARTICIPANT FLOW:
Groups:
- Cultivated Autologous Limbal Epithelial Cell (CALEC) Graft: Participants had a corneal biopsy in their non-diseased eye. A graft was manufactured for transplant using limbal epithelial cells, and transplanted into the diseased eye (CALEC transplant).
- Control Conjunctival Limbal Autograft (CLAU): Participants who were randomized to receive Conjunctival limbal autograft (CLAU) - Prior to this arm being ended. We dropped the control arm, which was IRB approved, due to low enrollment.
Period: Overall Study
Arm/Group | Cultivated Autologous Limbal Epithelial Cell (CALEC) Graft | Control Conjunctival Limbal Autograft (CLAU)
Started | 16 | 1
Completed | 14 | 1
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Failed Biopsy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants receiving a CALEC transplant, or the standard of care treatment (CLAU)
Groups:
- CALEC: Participants undergoing a biopsy with CALEC
- CLAU (Control): Participant(s) undergoing a biopsy with CLAU
- Total: Total of all reporting groups
Arm/Group | CALEC | CLAU (Control) | Total
Number analyzed (Participants) | 14 | 1 | 15
Age, Continuous [Median (Full Range); unit: Years] | 42.0 [24.0 to 78.0] | 53.0 [53.0 to 53.0] | 46.0 [24.0 to 78.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 13 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 1 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 14 | 1 | 15
Epithelial Integrity [Count of Participants; unit: Participants] — Number of Participants at Baseline with Epithelial Defect Surface Area
  Participants | 4 | 0 | 4
Epithelial Integrity [Median (Full Range); unit: units on a scale] — Corneal Surface Staining (NEI Grade Scale of 0 - 15) based on clinical assessments, where 0 us normal, and 15 is severe.
  units on a scale | 15.0 [10.0 to 15.0] | 10.0 [10.0 to 10.0] | 15.0 [10.0 to 15.0]
Neovascularization [Median (Full Range); unit: Neovascular Area (% of total area)] | 7.5 [0.5 to 24.2] | 3.6 [3.6 to 3.6] | 7.2 [0.5 to 24.2]
Ocular Surface Disease Index Score [Median (Full Range); unit: units on a scale] — The Ocular Surface Disease Index (OSDI) Score is scaled in the following:
  Normal: 0-12 points Mild: 13-22 points Moderate: 23-32 points Severe: 33-100 points
  units on a scale | 40.6 [6.8 to 100.0] | 95.5 [95.5 to 95.5] | 41.7 [6.8 to 100.0]
Symptom Assessment in Dry Eye Score [Median (Full Range); unit: units on a scale] — The Symptom Assessment in Dry Eye Score (SANDE) is scored and calculated by 0 which is normal, and 100 is Severe
  units on a scale | 35.4 [6.5 to 82.0] | 72.7 [72.7 to 72.7] | 39.1 [6.5 to 82.0]

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Events of Interest
Description: The occurrence of the following adverse events at any time during the 18 months of follow-up in the recipient eye will serve as the primary safety events of interest.
  1. Ocular Infection (defined as endophthalmitis or microbial keratitis [bacterial, fungal, parasitic]:
  2. Corneal Perforation
  3. Graft Detachment ≥50%
Time Frame: 18 Months
Population: All participants receiving a CALEC transplant or CLAU transplant.
Measure: Count of Participants; unit: Participants
Groups:
- CALEC: Participants undergoing a biopsy
- CLAU (Control): Participants undergoing CLAU procedure.
Arm/Group | CALEC | CLAU (Control)
Number analyzed (Participants) | 14 | 1
Participants
  Number of Participants with Ocular Infections | 1 | 0
  Number of Participants with Corneal Perforations | 0 | 0
  Number of Participants with Graft Detachments | 0 | 0

2. Primary Outcome: Manufacturing Feasibility Measures
Description: Each biopsy attempt will be classified as a "feasibility success" if it produced at least one construct that met all of the Quality Control (QC) release criteria. Manufacturing feasibility will be evaluate on a biopsy level (denominator is the total number of biopsies).The number and percentage of biopsy attempts resulting in a feasibility success will be calculated.
Time Frame: 18 Months
Population: Total number of biopsies performed. Fourteen of 16 biopsies (in 15 participants) resulted in a manufacturing success. Two failures occurred in the initial recruitment phase. One of the participant, had a second biopsy and successful transplant; the other elected not to return.
Measure: Number; unit: Biopsies
Units Other Than Participants: Biopsies
Arm/Group | CALEC
Number analyzed (Participants) | 15
Number analyzed (Biopsies) | 16
Biopsies | 14

3. Secondary Outcome: Measure of Transplant Efficacy
Description: The primary efficacy outcome will be a binary "Complete Success" of the graft defined as improvement in corneal surface integrity
Time Frame: 18 Months
Population: All participants undergoing a corneal biopsy. The total number of biopsy attempts are summarized.
Measure: Count of Participants; unit: Participants
Groups:
- CALEC: All participants undergoing a corneal biopsy. The total number of biopsy attempts are summarized.
- CLAU: All participants undergoing CLAU procedure. Total number of biopsy attempted are summarized.
Arm/Group | CALEC | CLAU
Number analyzed (Participants) | 14 | 1
Participants
  Complete Success : 3 Months Post Transplant | 7 | 1
  Complete Success : 12 Months Post Transplant | 11 | 0
  Complete Success : 18 Months Post Transplant | 10 | 1

ADVERSE EVENTS:
Time Frame: 18 Months
Description: Adverse Events Occurring in the Recipient Eye. Adverse Events Occurring in the Donor Eye. Systemic Adverse Events.
Groups:
- CALEC: Participants had a corneal biopsy in their non-diseased eye. A graft was manufactured for transplant using limbal epithelial cells and transplanted into the diseased eye (CALEC transplant)
- CLAU: Participants had a corneal biopsy in their non-disease eye, and transplanted into the the diseased eye.
Arm/Group | CALEC | CLAU
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/1
Other Adverse Events (participants affected / at risk) | 16/16 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CALEC (N=16) | CLAU (N=1)
Vomiting (Gastrointestinal disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CALEC (N=16) | CLAU (N=1)
Allergic Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Anterior Chamber Flare (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Blepharitis (Eyelid Irritation) (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Conjunctival Hyperemia (Eye disorders) | 12 (18) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Conjunctival Injection (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Corneal Bleeding (Eye disorders) | 9 (9) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Corneal Edema (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Corneal Epithelium Defect (Eye disorders) | 14 (38) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Corneal Neovascularization (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Dry Eye (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Ecchymosis - Skin (Eye disorders) | 3 (3) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Acne (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Discharge (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Infection NOS (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Irritation (Eye disorders) | 0 (0) | 1 (1) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Itching (Eye disorders) | 3 (3) | 1 (1) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Pain (Eye disorders) | 12 (17) | 1 (1) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Redness (Eye disorders) | 4 (5) | 1 (2) — Ocular Adverse Events Occurring in the Recipient Eye
Eye Tearing (Eye disorders) | 8 (8) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Eyelid Disorder (Eye disorders) | 1 (1) | 1 (1) — Ocular Adverse Events Occurring in the Recipient Eye
Foreign Body Sensation (Eye disorders) | 4 (5) | 1 (1) — Ocular Adverse Events Occurring in the Recipient Eye
Intraocular Pressure Increased (Eye disorders) | 3 (4) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Persistent Corneal Epithelial Defect (Eye disorders) | 5 (6) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Photophobia (Eye disorders) | 7 (10) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Sensitivity to Light (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Soreness in Eyes (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Recipient Eye
Subconjunctival Hemorrhage (Eye disorders) | 12 (12) | 1 (1) — Ocular Adverse Events Occurring in the Recipient Eye
Blurry Vision (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Conjunctival Disorder (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Conjunctival Hyperemia (Eye disorders) | 10 (10) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Corneal Edema (Eye disorders) | 7 (7) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Corneal Epithelium Defect (Eye disorders) | 15 (15) | 1 (2) — Ocular Adverse Events Occurring in the Donor Eye
Corneal Haze (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Corneal Neovascularization (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Ecchymosis - Skin (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Eye Irritation (Eye disorders) | 1 (1) | 1 (1) — Ocular Adverse Events Occurring in the Donor Eye
Eye Itching (Eye disorders) | 1 (1) | 1 (1) — Ocular Adverse Events Occurring in the Donor Eye
Eye Pain (Eye disorders) | 10 (10) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Eye Redness (Eye disorders) | 0 (0) | 1 (1) — Ocular Adverse Events Occurring in the Donor Eye
Eye Tearing (Eye disorders) | 5 (5) | 1 (1) — Ocular Adverse Events Occurring in the Donor Eye
Eyelid Margin Crusting (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Foreign Body Sensation in Eyes (Eye disorders) | 2 (2) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Hazy Vision (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Subconjunctival Hemorrhage (Eye disorders) | 11 (11) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Subconjunctival/Conjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0) — Ocular Adverse Events Occurring in the Donor Eye
Bruise (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Systemic Adverse Events
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Systemic Adverse Events
Fatigue (General disorders) | 0 (0) | 1 (1) — Systemic Adverse Events
Fever (General disorders) | 1 (1) | 0 (0) — Systemic Adverse Events
Foot Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Systemic Adverse Events
Headache (Nervous system disorders) | 9 (11) | 1 (1) — Systemic Adverse Events
Migrane Headache (Nervous system disorders) | 1 (1) | 0 (0) — Systemic Adverse Events
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Systemic Adverse Events
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Systemic Adverse Events
Streptococcal Sore (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Systemic Adverse Events
Toothache (General disorders) | 1 (1) | 0 (0) — Systemic Adverse Events
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Systemic Adverse Events
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Systemic Adverse Events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02592330/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT02592330/SAP_002.pdf
  • Informed Consent Form (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT02592330/ICF_003.pdf